CLINICAL TRIAL: NCT00307840
Title: Initial Dosing of Paricalcitol Based on iPTH Parathyroid Hormone Levels in Hemodialysis Patients With Secondary Hyperparathyroidism
Brief Title: Initial Dosing of Paricalcitol in Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Papageorgiou General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48/4-2-2005
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-03-28 (Estimated); Status verified 2005-08

CONDITIONS: Secondary Hyperparathyroidism
Keywords: hemodialysis; secondary hyperparathyroidism; hypercalcemia; hyperphosphatemia; vitamin D
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hypercalcemia; Hyperphosphatemia | interventions — paricalcitol

INTERVENTIONS:
Drug: paricalcitol

SUMMARY:
The purpose of this study was to compare two different initial dosing schemes for the administration of paricalcitol in hemodialysis patients with secondary hyperparathyroidism: the already in use iPTH/80 scheme, and an iPTH/120 scheme, which corresponds to the immediately lower dose, based on current instructions on paricalcitol dose adjustment. We studied the effectiveness of the two dosing schemes in achieving a target iPTH level (150 - 300 pg/mL)

DETAILED DESCRIPTION:
Adjustment of the initial dose of paricalcitol, in hemodialysis patients with secondary hyperparathyroidism (sHPT), on the basis of severity of sHPT is generally preferred in current practice. Whether the proposed dose, based on the formula baseline intact parathyroid hormone (iPTH [pg/mL]) divided by 80, is the most appropriate has not been adequately assessed. A trial comparing the iPTH/80 dose to the immediately lower iPTH/120 dose was undertaken. We studied the ability of the two different dosing schemes to control iPTH levels within a desired range between 150 and 300 pg/mL, as well as the frequency of iPTH over-suppression (< 150 pg/mL) in the two groups (iPTH/80 and iPTH/120).

ELIGIBILITY:
Inclusion Criteria:-maintenance hemodialysis therapy (3 sessions per week) for at least 3 months; iPTH between 300 and 900 pg/mL; age > 18 years; normal serum calcium concentration (8.1 - 10.4 mg/dL); Ca x P product less than 70; no vitamin D metabolite replacement therapy for at least one month prior to the enrollment; aluminum levels lower than 60 μg/L.

-

Exclusion Criteria:administration of calcitonin, disphosphonates or corticosteroids; presence of a clinically serious medical condition; previous parathyroidectomy; active malignancy.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Study Completion 2005-07

PRIMARY OUTCOMES:
The primary outcome was the achievement of desired iPTH levels (150 - 300 pg/mL) in the two groups (iPTH/80 and iPTH/120).

SECONDARY OUTCOMES:
The frequency of over-suppression of iPTH (< 150 pg/mL) was the secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Mitsopoulos, MD, Principal Investigator — Papageorgiou General Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Martin KJ, Gonzalez E, Lindberg JS, Taccetta C, Amdahl M, Malhotra K, Llach F. Paricalcitol dosing according to body weight or severity of hyperparathyroidism: a double-blind, multicenter, randomized study. Am J Kidney Dis. 2001 Nov;38(5 Suppl 5):S57-63. doi: 10.1053/ajkd.2001.28112. PMID 11689389